CLINICAL TRIAL: NCT04135313
Title: Induction and Consolidation Chemotherapy in Locally Advanced Rectal Cancer Patients With Circumferential Resection Margin Involvement: a Multicenter Prospective Randomized Phase III Clinical Trial
Brief Title: Induction and Consolidation Chemotherapy in Patients With Locally Advanced CRM-positive Rectal Cancer
Acronym: RuCorT-03
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Sergey Gordeyev, Principal Investigator, Consultant surgeon, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuCorT-03
Record Dates: First submitted 2019-10-20; First posted 2019-10-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Rectal Neoplasms Malignant; Rectum Carcinoma; Rectal Cancer
Keywords: rectal cancer; induction chemotherapy; consolidation chemotherapy; neoadjuvant chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy (Experimental): Patients receive 2 cycles of induction CapOx (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 per os bid days 1-14) chemotherapy, followed by chemoradiotherapy (54 Gy in 2 Gy fractions with concomitant capecitabine 825 mg/m2 per os bid on radiation days), then 2 cycles of consolidation CapOx chemotherapy, surgery (10-12 weeks following chemoradiotherapy) and 2 cycles of adjuvant CapOx chemotherapy
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy; Procedure: Rectal cancer surgery
- Chemoradiotherpy (Active Comparator): Patients receive 54 Gy pelvic chemoradiotherapy in 2 Gy fractions with capecitabine 825 mg/m2 bid per os on radiation days and then surgery following 10-12 weeks. After surgery patients receive 6 cycles of adjuvant CapOx chemotherapy.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy; Procedure: Rectal cancer surgery

INTERVENTIONS:
Drug: Capecitabine — 2000 mg/m2, bid, per os, days 1-14
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m2 iv day 1
Drug: Capecitabine — 825 mg/m2, bid, per os, only on days of radiation (Monday through Friday)
  Other Names: Xeloda
Radiation: Radiotherapy — Pelvic radiotherapy dose: 44 Gy on regional nodes, 54 Gy on primary tumor in 2 Gy fractions
Procedure: Rectal cancer surgery — Laparoscopic or open total mesorectal excision or extralevator abdominoperineal resection

SUMMARY:
The purpose of this study is to determine whether the addition of 2 cycles of induction CapOx chemotherapy and 2 cycles of consolidation CapOx chemotherapy to standard chemoradiation improves 3-year disease-free survival in patients with locally advanced CRM"+" mid and low rectal cancer.

DETAILED DESCRIPTION:
This trial aims to investigate the efficacy of adding neoadjuvant induction and consolidation chemotherapy compared to standard chemoradiotherapy in locally advanced rectal cancer patients with circumferential resection margin involvement. This is a prospective multicenter open-label randomized phase III clinical trial. Patients will be randomized using an online randomization system to receive either 2 cycles of induction CapOx (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 per os bid days 1-14) chemotherapy, followed by chemoradiotherapy (54 Gy in 2 Gy fractions with concomitant capecitabine 825 mg/m2 per os bid on radiation days), then 2 cycles of consolidation CapOx chemotherapy, surgery (10-12 weeks following chemoradiotherapy) and 2 cycles of adjuvant CapOx chemotherapy OR chemoradiotherapy (54 Gy in 2 Gy fractions with concomitant capecitabine 825 mg/m2 per os bid on radiation days), surgery (10-12 weeks following chemoradiotherapy) and 6 cycles of adjuvant CapOx chemotherapy. A stratification will be performed based on N stage, tumor location in the middle or low rectum and clinical center. Patients with middle or low rectal cancer without distant metastases, with involved circumferential resection margin (based on pretreatment MRI) will be included.

The target accrual is 270 patients in each treatment arm (including 10% potential data loss) based on potential benefit of 12% 3-yr disease-free survival (60% vs 72%), α=0,05, power 80% in the experimental arm. An interim analysis is planned after 50% of the patients will reach a 3-year followup. Pelvic Magnetic Resonance Imaging (MRI) is performed in all patients for staging before and after neoadjuvant chemotherapy and before surgery. Pelvic MRI is subject to central review. Conduction of this study and data collection are controlled by a local institutional board.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically verified colon rectal adenocarcinoma 0-10 cm above the anal verge
* No distant metastases
* Circumferential resection margin (CRM) involvement (based on pelvic MRI)
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Haemoglobin (HGB) > 90 g/L
* Platelet Count (PLT) > 120x10*9/L
* Serum creatinine < 150 µmol/L
* Total bilirubin < 25 µmol/L

Exclusion Criteria:

* inability to obtain informed consent
* distant metastases
* cT2N0M0 rectal cancer
* synchronous or metachronous tumors
* previous chemotherapy or radiotherapy
* clinically significant cardiovascular disorders (myocardial infarction < 6 months before visit, stroke < < 6 months before visit, instable angina < 3 months before visit, arrhythmia, uncontrolled hypertension > 160/100 mm hg
* clinically significant neurological disorders
* previous neuropathy 2 or higher
* current infection or heavy systemic disease
* pregnancy, breastfeeding
* ulcerative colitis
* individual intolerance to treatment components
* proven dihydropyrimidine dehydrogenase (DPD) deficiency
* participation in other clinical trials
* psychiatric disorders, which render patient unable to follow instructions or understand his/her condition
* technical inability to perform pelvic MRI
* inability of long-term followup of the patient
* HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Adjuvant chemotherapy compliance | 6 months
  Proportion of patients who receive a complete course of adjuvant chemotherapy
Acute chemotherapy toxicity | 6 months
  Toxicity measured according to NCI-CTCAE v.5.0
pathologic complete response rate (pCR) | 1 month
local recurrence rate | 3 years
3-year overall survival | 3 years
Operative morbidity | 30 days
  Morbidity measured according to Clavien-Dindo classification
Preoperative tumor-associated complications rate | 6 months
  The rate of tumor-associated complications (bowel obstruction, bleeding etc) during neoadjuvant chemotherapy
Sphincter preservation rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Zaman Z Mamedli, PhD, Principal Investigator — N.N.Blokhin Russian Cancer Research Center
Locations (1):
- N.N.Blokhin Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No